CLINICAL TRIAL: NCT00211835
Title: Treatment of Post-TBI Depression - A Randomized Clinical Trial
Brief Title: Treatment of Post-TBI Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCO 04-0782; H133B040033; NCT00233116 (obsolete NCT alias)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2013-09

CONDITIONS: Traumatic Brain Injury; Depression
Keywords: TBI; traumatic brain injury; depression; cognitive behavioral therapy; supportive psychotherapy; psychotherapy
MeSH Terms: conditions — Brain Injuries, Traumatic; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Arm 1 (Experimental): Individual psychotherapy focused on identifying and correcting maladaptive cognitions and behaviors with the goal of improving mood. The intervention has adapted CBT specifically to address cognitive deficits associated with TBI, which compound the cognitive distortions typical of depression. CBT therapists embed compensatory strategies within treatment sessions to address cognitive limitations of each participant.
  Interventions: Behavioral: Cognitive behavioral therapy
- Treatment Arm 2 (Experimental): A client-centered individual psychotherapy treatment approach designed to address depressive disorders commonly experienced by individuals following a TBI. In line with traditional supportive psychotherapy approaches, the objective of SPT is to improve the individual's ability to deal with problems of daily living more effectively through problem identification, praise, reassurance, encouragement, psychoeducation, advice, anticipatory guidance, and expanding awareness.
  Interventions: Behavioral: Supportive psychotherapy

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy — Individual psychotherapy focused on identifying and correcting maladaptive cognitions and behaviors with the goal of improving mood. The intervention has adapted CBT specifically to address cognitive deficits associated with TBI, which compound the cognitive distortions typical of depression. CBT therapists embed compensatory strategies within treatment sessions to address cognitive limitations of each participant.
  Arms: Treatment Arm 1
Behavioral: Supportive psychotherapy — A client-centered individual psychotherapy treatment approach designed to address depressive disorders commonly experienced by individuals following a TBI. In line with traditional supportive psychotherapy approaches, the objective of SPT is to improve the individual's ability to deal with problems of daily living more effectively through problem identification, praise, reassurance, encouragement, psychoeducation, advice, anticipatory guidance, and expanding awareness.
  Arms: Treatment Arm 2

SUMMARY:
Randomized clinical trial that compares the effects of cognitive behavioral therapy (CBT) and supportive psychotherapy for depression. Short- and long-term outcomes will be evaluated in terms of changes in mood (primarily depression and anxiety), participation in activities and life satisfaction.

DETAILED DESCRIPTION:
Goals Demonstrate the efficacy of cognitive behavioral therapy (CBT), both immediately after treatment and in the long term, in alleviating post-TBI depression.

Examine the relationship between improved mood, participation, and life satisfaction.

Implement exploratory analyses of the relationships between person and injury characteristics and outcomes of treatment.

Maximize potential application to clinical practice by:

Implementing the treatment in a clinical context so that its utility is demonstrated in a setting that maximizes ecological validity, and Creating and disseminating a manual detailing CBT treatment. This study is a randomized clinical trial that compares two treatment conditions: CBT and supportive psychotherapy (SPT). CBT has been shown to be effective in diverse studies. In this study, CBT has been shaped to be used specifically with people with typical post-TBI cognitive challenges. All participants will be given an opportunity to immediately receive a randomly assigned psychotherapy intervention to potentially enhance coping. Both CBT and SPT will involve 16 sessions of individual treatment. The initial session will be 90 minutes, with remaining sessions 50 minutes. In both treatments, participants will be seen for three months, with sessions twice weekly for the first month and once a week subsequently. The research assistants who will administer pre- and postintervention evaluation instruments will be blind to each participant's randomly assigned treatment condition. Evaluation instruments will be administered at baseline and at three points of follow-up: one week, six months, and one year after treatment. A detailed manual describing treatment methods will be developed based on the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Being at least 18years old
* Having a TBI as a result of a blow to the head followed by a loss of consciousness or period of being dazed and confused or a period of post traumatic amnesia or clinical signs of altered neurological function; this information must be medically documented (e.g., emergency medical record, hospital record, neuroradiological report, or neurological exam or record of physician's visit within 24 hours of injury)
* Being at least 6 months post injury
* Being English-speaking
* Having residential telephone service
* Living within 1.5 hours of New York City
* Having at least a sixth-grade reading level
* Meeting DSM-IV criteria for a current depressive mood disorder
* Not being in psychotherapy and being willing to abstain from seeking psychotherapy during the course of participation
* Being willing to complete questionnaires and interviews about mood, thinking skills, community participation and life satisfaction
* Agreeing to participate, verified by completion of informed consent and HIPAA documents.
* Individuals who meet criteria and are currently using prescribed mood medications will be included in the study if dosage has been stable for sixty days.

Exclusion Criteria:

* Pre-existing neurological disorder, including brain injury from an etiology other than trauma
* History of mental retardation
* Lack of capacity to sign informed consent
* Taking antidepressant medications for less than six months
* Having any changes in antidepressant medications in the last six months
* History of current or past psychosis or mania
* Current substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2005-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Remission of depression (DSM-IV diagnosis no longer met) | baseline
Remission of depression (DSM-IV diagnosis no longer met) | one week after treatment completion
Remission of depression (DSM-IV diagnosis no longer met) | six months after treatment completion
Remission of depression (DSM-IV diagnosis no longer met) | one year after treatment completion

SECONDARY OUTCOMES:
Increased participation (Participation Objective, Participation Subjective) | baseline
Improved quality of life (Life-3). | baseline
Increased participation (Participation Objective, Participation Subjective) | one week after treatment completion
Increased participation (Participation Objective, Participation Subjective) | six months after treatment completion
Increased participation (Participation Objective, Participation Subjective) | one year after treatment completion
Improved quality of life (Life-3). | one week after treatment completion
Improved quality of life (Life-3). | six months after treatment completion
Improved quality of life (Life-3). | one year after treatment completion

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Gordon, Ph.D., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Derived] Ashman T, Cantor JB, Tsaousides T, Spielman L, Gordon W. Comparison of cognitive behavioral therapy and supportive psychotherapy for the treatment of depression following traumatic brain injury: a randomized controlled trial. J Head Trauma Rehabil. 2014 Nov-Dec;29(6):467-78. doi: 10.1097/HTR.0000000000000098. PMID 25370439